CLINICAL TRIAL: NCT05724823
Title: Assessing a Telehealth Seated Exercise Program on Post-stroke Balance and Mobility: a Mixed-method Design
Brief Title: Virtual Physical Activity Seated Exercise - Phase 2
Acronym: V-PASE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Michael Smith Foundation for Health Research (Other)
Responsible Party: Principal Investigator, Janice Eng, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H22-02549
Record Dates: First submitted 2023-01-17; First posted 2023-02-13 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Chronic Stroke; Stroke, Ischemic; Stroke Hemorrhagic
Keywords: Stroke; Seated Exercise; Balance; Mobility; Cardiometabolic health; Randomized Controlled Trial
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 10-week group (Experimental): Will receive a 10-week seated exercise program, occurring 3 times per week. Sessions will be 60 minutes in duration.
  Interventions: Other: Virtual Physical Activity Seated Exercises (V-PASE)
- Delayed 2-week group (Boot Camp) (No Intervention): The Boot Camp group will complete a 2-week seated exercise program following the 10-week active trial period.

INTERVENTIONS:
Other: Virtual Physical Activity Seated Exercises (V-PASE) — The seated exercise program includes a variety of upper and lower limb strengthening, core strengthening, agility (fast arm and leg movements), and flexibility exercises. Participants will be supervised during each session thru videoconferencing by a trained instructor.
  Arms: 10-week group

SUMMARY:
This study will determine the acceptability of delivering seated exercises online and if seated exercises can improve balance, mobility, quality of life, and cardiometabolic health in those living with a stroke related mobility impairment.

Participants will be allocated to either a 10-week seated exercise program or a delayed 2-week Boot Camp program. All seated exercises sessions and assessments will be conducted virtually.

DETAILED DESCRIPTION:
The study will be a virtual 10-week multi-site, assessor-blinded, randomized controlled trial with an embedded qualitative component. The study will be conducted in real time using secure videoconferencing software (Zoom). Participants will be randomized 1:1 to a 10-week Seated Exercise group or a delayed 2-week Seated Exercise Group (Boot Camp). Seated exercise sessions will be delivered and supervised by a trained instructor.

Participants will use their own computer, laptop, or tablet for the zoom sessions. No Zoom sessions will be recorded. Caregivers will be invited to attend each exercise session to provide support and assistance but are not obliged to attend. A caregiver, friend, or family member will be required for each assessment to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following inclusion criteria:

* Adult (as defined by Province)
* Chronic stroke (more than 6 months post-stroke)
* Ability to stand up from a chair
* Mobility impairment of lower extremity (requires a walking aid, with or without close supervision)
* Able to safely engage in exercise and tolerate 60 minutes of exercises
* Able to communicate in English
* Have access to a tablet, computer, or laptop with internet and email access

Exclusion Criteria:

Participants will be excluded if they meet any of the following criteria:

* Participating in formal exercise or rehabilitation activities
* Participating in > 30 minutes/day of physical activity (moderate intensity)
* Participating in another study that may affect outcomes to this study
* Severe loss of vision, hearing, speech (including aphasia) or cognition that would preclude use of a computer/tablet and communication over videoconference software
* A serious comorbid condition (eg., amputation, Parkinson's disease, active cancer)
* Clinically diagnosed with acute/chronic illness or other condition which has known physical activity contraindications or limits their ability to complete each experimental condition (i.e., chronic low back pain aggravated by prolonged sitting)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
30 Second Sit-to-Stand | Immediately post-intervention (following 10-week trial)
  Assessment of balance and lower extremity strength.

SECONDARY OUTCOMES:
Timed Up and Go | Immediately post-intervention, and retention (2-months post-intervention)
  Participants stand up from a chair, walk 3 metres, turn around and then sit back down. The TUG assesses balance, mobility and turning ability
Tandem Stance | Immediately post-intervention, and retention (2-months post-intervention)
  Measures balance in standing as reported in the Short Physical Performance Battery Protocol
Modified Telehealth Fugl-Meyer | Immediately post-intervention, and retention (2-months post-intervention)
  The modified virtual Fugl-Meyer assess lower extremity impairments in those with stroke
Stroke Impact Scale | Immediately post-intervention, and retention (2-months post-intervention)
  A self-reported measure of stroke-related disability. There are 8 domains with each item rated using a 5-point Likert scale, where lower scores mean greater difficulty to complete the item.
Activities-Specific Balance Confidence (ABC) | Immediately post-intervention, and retention (2-months post-intervention)
  The ABC scale is a 16-item questionnaire where a participant rates their confidence in performing activities from 0% to 100% (higher percentages indicate greater self-efficacy).
Fatigue Severity Scale | Immediately post-intervention, and retention (2-months post-intervention)
  Questionnaire assessing the impact of fatigue on daily tasks and activities. There are 9 questions, each scored from 1 to 7 (1 = strongly disagree; 7 = strong agreement).
Quality of Life (EQ-5D-5L) | Immediately post-intervention, and retention (2-months post-intervention)
  The EQ-5D-5L assess self-care, mobility, depression/anxiety, pain, and usual activities. Each is scored with 5 levels (1=no problems, 5=major problems). Overall health on the day is scored from 0% (worst health) to 100% (best health).
Patient Health Questionnaire-4 (PHQ-4) | Immediately post-intervention, and retention (2-months post-intervention)
  The PHQ-4 focuses on depression and anxiety. Questions are scored from 0 to 3 (0=not at all; 3 = Nearly every day).
Montreal Cognitive Assessment scale (MoCA-BLIND) | Immediately post-intervention, and retention (2-months post-intervention)
  The MoCA-BLIND assess six different cognitive domains (excludes visual stimulus) over the phone: memory, attention, language, abstraction, delayed recall, and orientation. The MoCA-BLIND is scored from 0-22 (22 = no cognitive impairments).
Lipid Profiles | Immediately post-intervention, and retention (2-months post-intervention)
  Blood samples will be collected following a 12-hour over-night fast
Fasting Glucose | Immediately post-intervention, and retention (2-months post-intervention)
  Blood samples will be collected following a 12-hour over-night fast
Glucose (HbA1c) | Immediately post-intervention, and retention (2-months post-intervention)
  Blood samples will be collected following a 12-hour over-night fast
30 Second Sit-to-Stand | Retention (2-months post-intervention)
  Assessment of balance and lower extremity strength.

OTHER OUTCOMES:
Feasibility Indicator: Compliance | Through study completion (approximately 10 weeks)
  Percentage of participants that attend exercise sessions.
Feasibility Indicator: Safety | Through study completion (approximately 10 weeks)
  Number of adverse events that occur during assessments or exercise sessions.

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - GF Strong Rehabilitation Centre, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Nova Scotia Health, Halifax, Nova Scotia
  - Western University, London, Ontario
  - University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mackie P, Ashe MC, Barclay R, Bayley MT, Donkers SJ, Fleet JL, Mortenson WB, Peters S, Pollock CL, Pooyania S, Quigley A, Sakakibara BM, Schneeberg A, Sheehy L, Stelling S, Yao J, Eng JJ. Transferability of a 10-week remotely delivered Virtual Physical Activity Seated Exercise (V-PASE) program on post-stroke functional mobility: study protocol for a multisite randomized controlled trial. Trials. 2026 Feb 6. doi: 10.1186/s13063-026-09523-8. Online ahead of print. PMID 41645237